CLINICAL TRIAL: NCT00132067
Title: A Phase II Evaluation of Vorinostat, (SAHA, NCI-Supplied Agent [NSC #701852]) in the Treatment of Persistent or Recurrent Epithelial Ovarian or Primary Peritoneal Carcinoma
Brief Title: Vorinostat in Treating Patients With Recurrent or Persistent Ovarian Epithelial or Primary Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02667; NCI-2012-02667 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG 0170H; CDR0000439489; GOG-0170H (Other: Gynecologic Oncology Group); GOG-0170H (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2005-08-16; First posted 2005-08-19 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Vorinostat

ARMS (1):
- Treatment (vorinostat) (Experimental): Patients receive oral vorinostat twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: vorinostat

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza

SUMMARY:
This phase II trial is studying how well vorinostat works in treating patients with recurrent or persistent ovarian epithelial or primary peritoneal cavity cancer. Drugs used in chemotherapy, such as vorinostat, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 6-month progression-free survival rate in patients with recurrent or persistent ovarian epithelial or primary peritoneal cavity cancer treated with vorinostat.

II. Determine the toxicity of this drug, in terms of the frequency and severity of adverse reactions in these patients.

SECONDARY OBJECTIVES:

I. Determine the clinical response rate (partial response and complete response) in patients treated with this drug.

II. Determine the duration of progression-free survival and overall survival of patients treated with this drug.

III. Determine the impact of prognostic variables (e.g., platinum sensitivity, performance status, and cellular histology) in patients treated with this drug.

OUTLINE: This is a nonrandomized, multicenter study.

Patients receive oral vorinostat twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-60 patients will be accrued for this study within approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal cavity cancer
* Recurrent or persistent disease

  * Disease progression during OR persistent disease after completion of 1 prior platinum-based chemotherapy regimen (containing carboplatin, cisplatin, or other organoplatinum compound) for primary disease

    * Initial treatment may have included high-dose, consolidation, noncytotoxic agents, or extended therapy administered after surgical or non-surgical assessment
    * Treatment-free interval after completion of platinum-based chemotherapy must have been < 12 months
* Measurable disease, defined as ≥ 1 unidimensionally measurable target* lesion ≥ 20 mm by conventional techniques (e.g., palpation, plain x-ray, CT scan, or MRI) OR ≥ 10 mm by spiral CT scan
* Not eligible for a higher priority GOG protocol (i.e., any active phase III GOG protocol for the same patient population)
* No known brain metastases
* Performance status - GOG 0-1
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Able to take oral medication
* No bowel obstruction
* No persistent vomiting
* No parenteral feeding
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 1 month after completion of study treatment
* No neuropathy (sensory and motor) > grade 1
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No active infection requiring antibiotics
* No psychiatric illness or social situation that would preclude study compliance
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to vorinostat
* No other uncontrolled illness
* At least 4 weeks since prior immunotherapy for the malignancy
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) for the malignancy and recovered
* No more than 2 prior cytotoxic chemotherapy regimens for recurrent or persistent disease
* No prior non-cytotoxic chemotherapy for recurrent or persistent disease, unless therapy was part of the primary treatment regimen
* No prior vorinostat
* At least 1 week since prior hormonal therapy for the malignancy
* Concurrent hormone replacement therapy allowed
* At least 4 weeks since prior radiotherapy for the malignancy and recovered
* No prior radiotherapy to > 25% of bone marrow
* At least 4 weeks since prior surgery for the malignancy and recovered
* At least 4 weeks since other prior therapy for the malignancy
* At least 30 days since prior and no concurrent valproic acid
* Concurrent oral anticoagulants (i.e., warfarin) allowed provided there is increased vigilance with respect to monitoring PT/INR for the first 2 courses of study therapy or if there are any signs of bleeding
* No prior anticancer therapy that would preclude study participation
* No concurrent combination anti-retroviral therapy for HIV-positive patients
* No other concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | At 6 months
  Time at risk will be assessed from the date of registration onto the study and include all eligible patients who receive any study treatment. An analysis of any potential treatment effect on PFS may be conducted against the historical controls provided in GOG 126 and GOG 146 using a proportional hazards model that includes histological cell type, performance status, and platinum sensitivity.
Toxicity as assessed by CTCAE v 3.0 | Up to 5 years after completion of study treatment

SECONDARY OUTCOMES:
Clinical response (partial and complete response) rate as according to RECIST s | Up to 5 years
Duration of PFS | From study entry until disease progression, death or date of last contact., assessed up to 5 years
Duration of survival | From entry into the study to death or the date of last contact, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susan Modesitt, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States